CLINICAL TRIAL: NCT07263802
Title: Evaluation of the Efficacy of GlycoDual on Postprandial Glycemic Control and Insulin Sensitivity in Subjects With Impaired Glucose Metabolism: a Randomized, Controlled, Double-blind Study
Brief Title: Effect of a Food Supplement on Glycemic Parameters in Patients With Impaired Glucose Metabolism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Giuseppe Derosa, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDUAL-2025-RCT01
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Impaired Fasting Glucose (IFG); Impaired Glucose Tolerance (Prediabetes)
Keywords: dysglycemia; Gymnema sylvestre; Zinc bisglycinate
MeSH Terms: conditions — Glucose Intolerance; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Patients taking nutraceutical
  Interventions: Dietary Supplement: GlycoDual
- Placebo (Placebo Comparator): Patients taking placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: GlycoDual — GlycoDual is a food supplement developed to control post-prandial glycemia and improve insulin sensitivity in subjects with impaired glucose metabolism. GlycoDual contains maqui berry, blueberry, cocoa (rich in anthocyanins and epicatechin), and chromium picolinate, aimed at modulating the immediate glycemic response through the inhibition of α-glucosidase, stimulation of glucose transport and insulin sensitization. It also contains Gymnema sylvestre and zinc bisglycinate, aimed at supporting insulin secretion and contributing to the long-term regulation of glycemia
  Arms: Intervention
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective will be to evaluate the efficacy of GlycoDual in reducing fasting plasma glucose (FPG) and post-prandial plasma glucose (PPG) levels compared to placebo after 90 days of treatment.

Secondary objectives are to estimate:

* the change of insulin sensitivity (HOMA-IR)
* the change of uricemia after 90 days of supplementation compared to placebo.

Safety objectives: Collection of the adverse events not related, related or possibly related to the study products.

DETAILED DESCRIPTION:
Mild dysglycemias, such as impaired fasting glucose (IFG) and impaired glucose tolerance (IGT), represent pre-diabetic conditions characterized by a subclinical impairment of insulin sensitivity and β-cell function. Early intervention in this phase can prevent or delay the progression to full-blown diabetes. In this context, the use of nutraceutical supplements with physiological activity on glucose metabolism represents a promising and well-tolerated approach, able to effectively modulate metabolic parameters, with a good safety profile. GlycoDual is a food supplement developed to control post-prandial glycemia and improve insulin sensitivity in subjects with impaired glucose metabolism. GlycoDual contains maqui berry, blueberry, cocoa (rich in anthocyanins and epicatechin), and chromium picolinate, aimed at modulating the immediate glycemic response through the inhibition of α-glucosidase, stimulation of glucose transport and insulin sensitization. It also contains Gymnema sylvestre and zinc bisglycinate, aimed at supporting insulin secretion and contributing to the long-term regulation of glycemia The primary objective will be to evaluate the efficacy of GlycoDual in reducing fasting plasma glucose (FPG) and post-prandial plasma glucose (PPG) levels compared to placebo after 90 days of treatment.

Secondary objectives are to estimate:

* the change of insulin sensitivity (HOMA-IR)
* the change of uricemia after 90 days of supplementation compared to placebo.

Safety objectives: Collection of the adverse events not related, related or possibly related to the study products.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) 25.0-29.9 kg/m2
* FPG levels between 100 and 125 mg/dl [IFG diagnosed after Oral Glucose Tolerance Test (OGTT)]
* HOMA-IR > 2.5
* subjects able to understand the informed consent and sign it before enrollment in the study

Exclusion Criteria:

* personal history of cardiovascular disease or equivalent risk factors
* obesity (BMI ≥ 30 kg/m²)
* taking hypoglycemic drugs or supplements that affect glycemic metabolism
* diabetes mellitus or IGT
* pregnancy or breastfeeding
* known thyroid, liver, kidney or muscle diseases
* any medical or surgical condition that makes patient compliance with the study protocol complex or inconsistent
* any known allergy or hypersensitivity to one or more components of the food supplement

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Effects on glycemia | 90 days
  evaluate the efficacy of GlycoDual in reducing fasting plasma glucose (FPG) and post-prandial plasma glucose (PPG) levels compared to placebo after 90 days of treatment.

SECONDARY OUTCOMES:
Change in Insulin sensitivity | 90 days
  The secondary objective will be to evaluate the efficacy of GlycoDual in reducing insulin sensitivity (HOMA-IR) levels compared to placebo after 90 days of treatment.
Change in uricemia | 90 days
  The secondary objective will be to evaluate the efficacy of GlycoDual in reducing uricemia levels compared to placebo after 90 days of treatment.

IPD SHARING:
Plan to Share IPD: No